CLINICAL TRIAL: NCT02400021
Title: Progesterone Supplementation for HIV-positive Pregnant Women on Anti-Retrovirals
Acronym: ProSPAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTNPT025
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prometrium (Experimental): Prometrium (progesterone capsules) intervention
  Interventions: Drug: Prometrium
- No treatment (No Intervention): no treatment arm

INTERVENTIONS:
Drug: Prometrium
  Other Names: progesterone capsules
  Arms: Prometrium

SUMMARY:
In pregnancy, cART is considered optimal for maternal health and for preventing the emergence of resistance that could compromise further care. In Canada, the majority of HIV-positive pregnant women receive a PI-based cART regimen. In the past, therapy was generally deferred until after the first trimester (if not required for maternal health) to minimize any unknown risk of teratogenicity. However, as treatment is now started earlier in HIV infection and as perinatal transmission rates are lowest in those with prolonged suppression of viral load during pregnancy, women are increasingly commencing cART either before conception or earlier in pregnancy.

Multiple reports and cohort studies provided data suggesting an association between PI-based cART use and preterm birth, low birth weight, and small for gestational age (SGA) babies, although conflicting data exist.

In the general population progesterone supplementation is widely used, is well tolerated, is considered safe, and is beneficial to prevent recurrent pre-term birth and increase birth weight. The investigators experimental findings suggest that PI use during pregnancy is associated with declines in progesterone levels that correlate with fetal growth, and that progesterone supplementation can improve PI-induced fetal growth restriction. The investigators preliminary findings in HIV+ pregnant women suggest that PI-use is associated with declines in progesterone levels, which correlate with birth weight percentile. Since HIV-positive women have higher rates of pre-term delivery and low birth weight that may be magnified by the use of PIs, then progesterone supplementation could be of benefit to neonatal health in the context of HIV-positive pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* On (stable) or initiating a cART regimen containing either ritonavir-boosted lopinavir (LPV/r), atazanavir (ATZ/r) or darunavir (DRV/r)
* Pregnant up to 24 weeks gestational age
* Singleton pregnancy
* 18 years or older
* Ability to give informed consent

Exclusion Criteria:

* Hypersensitivity or allergy to soya or peanut (non-active ingredient supplement in Prometrium)
* Contraindications to intravaginal progesterone use including:

  * documented hypersensitivity to Prometrium
  * active or history of breast cancer,
  * active or history of arterial thromboembolitic disease (e.g. stroke, myocardial infarction, coronary heart disease)
  * active or history of venous thromboembolism (e.g. deep venous thrombosis or pulmonary embolism) or active thrombophlebitis
  * any prior neoplasia, except for skin
  * abnormal vaginal bleeding
* Known lethal fetal anomaly
* Any contraindication to continuation of pregnancy
* Inability to communicate in English
* Prior participation in this trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Total enrollment / eligible population per year | 12 months
  Qualitative information on the reasons to decline participation will be collected and summarized. Reasons for non-enrolling questionnaire will be used.

SECONDARY OUTCOMES:
Safety of progesterone supplementation during pregnancy for HIV-positive women. | 40 weeks
  The number of Grade 3 or 4 AE in the ITT vs. comparator group. The number of Grade 1 or 2 AE in the ITT vs. comparator group. AE questionnaire.
Acceptability of progesterone supplementation during pregnancy for HIV+ women. | 40 weeks
  Assessed in the ITT group. Acceptability based on experience with medication questionnaire. Screening questionnaire (acceptability of being recruited to no treatment arm)
Compliance of progesterone supplementation. Assessed in the ITT group. | 40 weeks
  Number of missed doses / total prescribed doses per patient. Compliance questionnaire
Barriers to adherence to progesterone supplementation. Assessed in the ITT group | 40 weeks
  Reasons for missed dose questionnaire. Reasons for missed appointment questionnaire

OTHER OUTCOMES:
Serum progesterone levels at GW25-28 and GW33-36, described by treatment group. | 28 weeks, 36 weeks
  SD and intra-patient correlation coefficient of trough serum progesterone levels will be calculated
Urine progesterone levels at GW25-28 and GW33-36, described by treatment group | 28 weeks, 36 weeks
  SD and intra-patient correlation coefficient will be calculated.
Distribution of birth weight, birth weight percentile, and gestational age at birth, compared by treatment group. | 40 weeks
  ITT and on-treatment analysis
Relationship between progesterone levels (serum or urine) at GW25-28 or GW33-36 and birth weight, birth weight percentile, and gestation age at birth. | 28 weeks, 36 weeks
  assessed with spearman's rank correlation
Serum/urine progesterone levels compared between women with and without an AE/SAE. | 40 weeks
Biomarker analysis | 40 weeks
  levels of sex steroids, angiogenic, vasoactive, and inflammatory factors, factors associated with placentation, placenta dysfunction, pre-term delivery and fetal growth restriction between treatment groups
Placenta morphology between treatment groups | 40 weeks
  Qualitative assessment performed blinded to the arm allocation and birth outcome
Progesterone supplementation effect on PI drug levels | 40 weeks
  trough PI drug levels in plasma collected from women in both tx groups at baseline and each study visit. changes in drug levels over time will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Walmsley, MD, Principal Investigator — Toronto General Research Institute, UHN; Kellie Murphy, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (5):
- Canada (5):
  - St. Joseph's Hospital, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Maple Leaf Medical Clinic, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Siou K, Walmsley SL, Murphy KE, Raboud J, Loutfy M, Yudin MH, Silverman M, Ladhani NN, Serghides L. Progesterone supplementation for HIV-positive pregnant women on protease inhibitor-based antiretroviral regimens (the ProSPAR study): a study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2016 Aug 12;2:49. doi: 10.1186/s40814-016-0087-6. eCollection 2016. PMID 27965866